CLINICAL TRIAL: NCT01671891
Title: Detection and Enumeration of Circulating Tumor Cells in Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, director of radiotherapy department in Fudan university shanghai cancer center, Fudan University
Other Study IDs: SCRC-NM-1001
Record Dates: First submitted 2012-07-19; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; circulating tumor cells; predict responses
MeSH Terms: conditions — Rectal Neoplasms; Neoplastic Cells, Circulating | interventions — Radiotherapy; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- rectal cancer with stage II-IV: rectal cancer with stage II-IV intervention: pelvic radiotherapy (45-55Gy) concurrent chemotherapy using capecitabine and oxaliplatin
  Interventions: Radiation: radiation therapy; Drug: capecitabine (625mg/m2,bid,d1-5 qw)and oxaliplatin (85mg/m2 d1 qw)

INTERVENTIONS:
Radiation: radiation therapy — 45-55Gy
Drug: capecitabine (625mg/m2,bid,d1-5 qw)and oxaliplatin (85mg/m2 d1 qw) — radiotherapy concurrent chemotherapy(capecitabine+oxaliplatin)
  Other Names: Xeloda

SUMMARY:
Rectal cancer is one of the most common malignant tumors in the world. However, there's also no reliable and sensitive method to monitor diseases and evaluate therapy responses till now. Circulating tumor cells, which could reflect tumor's status correctly and reliably, may be a promising method in this field. This study is to investigate the role of circulating tumor cells in evaluating and predicting the responses of chemoradiotherapy in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified rectal carcinoma
* Locally advanced tumor (cT3-4 and/or N+ by transrectal ultrasound and/or pelvic magnetic resonance imaging)
* the distance from anal verge <= 12cm
* with or without metastasis
* Age 18-75 years old
* ECOG PS 0-2
* No previous chemotherapy or radiotherapy for rectal carcinoma
* Written informed consent

Exclusion Criteria:

* no histologically verified rectal carcinoma
* rectal cancer with stage I
* distance from verge >12cm
* age <=18 or >=75 years old
* performed previously chemotherapy or radiotherapy
* infection diseases within three months
* serious other diseases
* no written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: rectal cancer diagnosed with stage II-IV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
circulating tumor cells level changes after radiotherapy | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
disease-free survival | 3 years
serum carcinoembryonic antigen (CEA) level | 3 years
pathological response (tumor regression grade)if surgery | 3 years
RECIST-based tumor response at 10 week after radiotherapy | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China, China

REFERENCES:
- See also: circulating tumor cells in colorectal cancer — http://www.ncbi.nlm.nih.gov/pubmed/22230943
- See also: Circulating tumors cells as biomarkers: progress toward biomarker qualification — http://www.ncbi.nlm.nih.gov/pubmed/22157288